CLINICAL TRIAL: NCT01738139
Title: A Phase I Trial of Ipilimumab (Immunotherapy) and Imatinib Mesylate (c-Kit Inhibitor) in Patients With Advanced Malignancies
Brief Title: Ipilimumab and Imatinib Mesylate in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0784; NCI-2018-01811 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0784 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Advanced Malignant Solid Neoplasm; C-KIT Tyrosine Kinase Protein Overexpression; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Gastrointestinal Stromal Tumor; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Unresectable Melanoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis; Melanoma | interventions — Imatinib Mesylate; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ipilimumab, imatinib mesylate) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1 and imatinib mesylate PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Imatinib Mesylate; Biological: Ipilimumab

INTERVENTIONS:
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy

SUMMARY:
This phase I trial studies the side effects and best dose of ipilimumab and imatinib mesylate in treating patients with solid tumors that have spread to other places in the body or cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving ipilimumab and imatinib mesylate may work better in treating patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity profile of intravenous ipilimumab (Yervoy) administered in combination with oral imatinib mesylate (GLEEVEC) for patients with advanced malignancies that are refractory to standard therapy, relapsed after standard therapy, or have no available standard therapy.

II. To determine the maximum toxic dose (MTD) and dose limiting toxicities (DLT) of ipilimumab and imatinib mesylate combination therapy.

SECONDARY OBJECTIVES:

I. To determine antitumor activity of ipilimumab and imatinib mesylate combination therapy.

II. To determine antitumor activity of ipilimumab and imatinib mesylate combination therapy in KIT confirmed solid tumors.

III. To evaluate the potential predictive role of tumor-associated immune biomarkers for therapy effectiveness.

IV. To evaluate the potential predictive role of therapy associated toxicities with antitumor activity.

OUTLINE: This is a dose-escalation study.

Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1 and imatinib mesylated orally (PO) twice daily (BID) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation study, patients must have histological confirmation of solid tumors that is metastatic or unresectable. For expansion cohorts, patients must have metastatic or unresectable gastrointestinal stromal tumor (GIST), melanoma, or uncategorized tumors with tumor biopsies that are positive for c-KIT mutations by polymerase chain reaction (PCR) or immunohistochemistry (IHC). For patients enrolled in the melanoma expansion cohort, only select KIT mutations will be eligible. Patients with mutations in exon 13 V654X, 14 T6701, 17 D816X and all exon 18 mutations will not be eligible for enrollment.
* Patients who have completed previous therapies 4-weeks prior to (or within 5 drug half lives) enrollment on study. Radiation therapy wash out period will be 2 weeks. This includes an exception of patients with metastatic GIST tumors who are taking maintenance imatinib mesylate therapy. These patients are allowed to remain on imatinib mesylate therapy up to enrollment in this study.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%).
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Total bilirubin < or = 2.0 mg/dL. (Does NOT apply to patients with Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal (patients with liver involvement will be allowed < or = 5.0 X institutional upper normal limit)
* Serum creatinine < 2.0 mg/dL
* Patients MUST have recovered from all treatment related toxicities to grade 1 National Center Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version [v] 4.0) in severity.
* Patients must be willing and able to review, understand, and provide written consent before starting therapy.
* Patients with histologically proven intracranial glioblastoma, gliosarcoma or anaplastic astrocytoma will be eligible. Patients must have shown unequivocal radiographic evidence for tumor progression by magnetic resonance imaging (MRI) scan. A scan should be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required.
* Patients in the expansion cohort must also agree to participate in the biomarker study. However, patients in the melanoma KIT positive mutant subgroup, patients must agree to participate in the biomarker study and biopsies.
* Patients must be willing to stay within 2 hours drive of MD Anderson Cancer Center whilst receiving Ipilimumab therapy. Patient must also agree to present to MD Anderson emergency center while on Ipilimumab therapy.

Exclusion Criteria:

* Autoimmune disease: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus or autoimmune vasculitis [e.g., Wegener's granulomatosis] are excluded from this study.
* History of acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation.
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events (AEs): e.g. a condition associated with frequent diarrhea or chronic skin conditions, recent surgery or colonic biopsy from which the patient has not recovered, or partial endocrine organ deficiencies.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Any non-oncology live vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab).
* Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids (when used in the management of cancers other than intracranial glioblastoma, gliosarcoma or anaplastic astrocytoma, or when used to treat non-cancer-related illnesses).
* Patients who do not agree to practice appropriate birth control methods while on therapy.
* Pregnant women are excluded from this study. Women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-02-19 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 7 years
Maximum tolerated dose (MTD) | 84 days
  MTD determined as the highest dose level with less than 2 patients with dose limiting toxicity (DLT) out of at least six patients in the cohort. DLT determined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Reilley MJ, Bailey A, Subbiah V, Janku F, Naing A, Falchook G, Karp D, Piha-Paul S, Tsimberidou A, Fu S, Lim J, Bean S, Bass A, Montez S, Vence L, Sharma P, Allison J, Meric-Bernstam F, Hong DS. Phase I clinical trial of combination imatinib and ipilimumab in patients with advanced malignancies. J Immunother Cancer. 2017 Apr 18;5:35. doi: 10.1186/s40425-017-0238-1. eCollection 2017. PMID 28428884
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org